CLINICAL TRIAL: NCT06335550
Title: Pilot Robotic Mastectomy in Singapore (PRoMiSing I) Study: First Safety and Feasibility Prospective Cohort Study in South East Asia
Brief Title: Surgical and Patient Reported Outcomes in Robotic Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changi General Hospital (Other)
Responsible Party: Principal Investigator, Mok Chi Wei, Principal Investigator; Clinical Assistant Professor, Changi General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021/2680
Record Dates: First submitted 2024-03-04; First posted 2024-03-28 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Minimally invasive breast surgery; endoscopic breast surgery; robotic breast surgery
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Robotic mastectomy (Other): All consecutive cases of robotic mastectomy over the study duration
  Interventions: Procedure: Robotic mastectomy

INTERVENTIONS:
Procedure: Robotic mastectomy — Robotic mastectomy with or without reconstruction

SUMMARY:
Conventional nipple and/or skin-sparing mastectomy (NSM/SSM) with or without immediate reconstruction is becoming one of the mainstream surgical treatment for breast cancer and risk reducing mastectomy in recent years. While this technique provides satisfactory oncologic and aesthetic outcomes, its disadvantages include skin flap and/or nipple-areolar complex (NAC) necrosis, NAC malposition/distortion as well as visible scar(s) on the breast.

In terms of technical aspects, NSM/SSM has its inherent challenges in view of limited incisions and thereby difficulties in dissection. Since 2015, a number of institutions worldwide had adopted a new technique of NSM/SSM using robotic surgical system. Institutional experiences worldwide demonstrated feasibility and safety of this technique coupled with improved patients' satisfactions.

To date, there is no center in Singapore or the region offering Robotic NSM/SSM (R-NSM/R-SSM). The authors believe that robotic mastectomy is a feasible and safe technique that can be utilized in our institution and it provides superior aesthetic outcomes with less morbidity and higher patient satisfaction if compared to conventional NSM/SSM.

The aim of this study is to conduct a single-arm prospective pilot study to investigate the safety and feasibility as well as learning curve of R-NSM/R-SSM.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 21-70, with invasive breast cancer, ductal carcinoma in situ (DCIS), Breast Cancer (BRCA) gene or other breast cancer genetic mutation carriers or high risk female patients who are otherwise candidates for conventional NSM/SSM will be eligible for the study. All suitable patients will be offered the option of R-NSM/ R-SSM.

For patients with breast cancer (invasive or DCIS), selection criteria include but not limited to:

1. Early breast cancer
2. Tumor size less than 5 cm
3. No evidence of lymph node metastases
4. No evidence of skin or chest wall invasion.

Exclusion Criteria:

1. Extensive axillary lymph node metastasis (Stage 3B or later)
2. Heavy smokers (>20 cigarettes a day)
3. High risk patient with severe and poorly controlled co-morbid conditions (include but not limited to diabetes, heart disease, renal failure or liver dysfunction)
4. Poor performance status or high risk for anaesthesia (ASA 3 and above)
5. Inflammatory or Locally Advanced Breast Cancer (with or without chest wall or skin invasion)

Ages: 21 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2022-11-24 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Surgical Outcomes - Operative parameters | Postoperative Day 0-1
  - Operative parameters (in terms of docking time/console time and total operative time - defined as time taken from axilla staging procedure, robot docking time, console time, closure and time taken for reconstruction, if applicable
Surgical Outcomes - Length of stay (days) | Postoperative 30 days
  - Length of stay (days)
Surgical Outcomes- 30-days morbidity/complications | Postoperative 30 days
  - 30-days morbidity/complications

SECONDARY OUTCOMES:
Oncologic outcomes | Postoperative 2 weeks until final histopathology results are available
  Short-term oncologic outcomes, such as positivity of margins
Learning curve | Postoperative up to 2 years throughout study recruitment
  Learning curve analysis using cumulative sum (CUSUM) method

CONTACTS AND LOCATIONS:
Overall Officials: Chi Wei Mok, Principal Investigator — Changi General Hospital
Locations (1):
- Changi General Hospital, Singapore, Singapore

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-07-05): https://cdn.clinicaltrials.gov/large-docs/50/NCT06335550/Prot_SAP_000.pdf
  • Informed Consent Form (2023-05-03): https://cdn.clinicaltrials.gov/large-docs/50/NCT06335550/ICF_001.pdf